CLINICAL TRIAL: NCT01328002
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Withdrawal Study to Evaluate the Safety, Tolerability, and Efficacy of Milnacipran in Pediatric Patients With Primary Fibromyalgia
Brief Title: Safety and Efficacy of Milnacipran in Pediatric Patients With Primary Fibromyalgia
Acronym: MyFi
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Cypress Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN-MD-14
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-03

CONDITIONS: Primary Fibromyalgia
Keywords: Fibromyalgia; Pediatric Fibromyalgia; Adolescent Fibromyalgia; milnacipran; Savella; loss of therapeutic response; Forest Research Institute; Pain; Fatigue; Serotonin Norepinephrine Reuptake Inhibitors; Randomized Withdrawal
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milnacipran (Experimental): oral administration, twice daily dosing
  Interventions: Drug: Milnacipran
- Placebo (Placebo Comparator): oral administration, twice daily dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — Maximum tolerated dose (50, 75, or 100 mg/day tablets) was determined during the open label phase of the study.
  Oral administration, twice daily dosing
  Other Names: Savella
  Arms: Milnacipran
Drug: Placebo — matching placebo tablets daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, efficacy, and pharmacokinetics of milnacipran in pediatric patients aged 13 to 17 years with primary fibromyalgia.

DETAILED DESCRIPTION:
* 8 weeks open-label treatment period with milnacipran.
* Followed by randomization to 8-weeks double blind treatment period for eligible patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary fibromyalgia
* 13-17 years of age
* To be eligible for screening, have average pain rating in the previous week of at least 3 but no more than 9 on an 11-point numeric rating scale
* To be eligible to enter into the open-label treatment period, have a 1-week mean of daily pain ratings of at least 3 but no more than 9 (11-point numeric rating scale) in the week before Baseline (Visit 2)
* To be eligible for randomization and entry into the double-blind treatment period, have a decrease of at least 50% in 1-week mean of daily pain ratings (11-point numeric rating scale) before Randomization (Visit 7) compared with the 1-week mean of daily pain ratings, in the week before Baseline (Visit 2)
* Unsatisfactory response to nonpharmacologic fibromyalgia treatment.

Exclusion Criteria:

* Severe psychiatric illness
* Severe renal impairment
* Evidence of active liver disease
* Pregnant or breastfeeding
* Significant risk of suicidality
* Unable, unwilling or inadvisable to discontinue prohibited medications
* History of alcohol abuse or drug abuse or dependence, within previous year
* Current systemic infection
* Autoimmune disease
* History of seizure disorder (other than febrile seizures)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2011-04-30 (Actual); Primary Completion 2012-08-31 (Actual); Study Completion 2012-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M D'Astoli, LPN, Study Director — Forest Laboratories
Locations (47):
- United States (47):
  - Forest Investigative Site 040, Birmingham, Alabama
  - Forest Investigative Site 068, Birmingham, Alabama
  - Forest Investigative Site 033, Bullhead City, Arizona
  - Forest Investigative Site 012, Fresno, California
  - Forest Investigative Site 045, Fresno, California
  - Forest Investigative Site 051, Fresno, California
  - Forest Investigative Site 035, Orange, California
  - Forest Investigative Site 053, Orange, California
  - Forest Investigative Site 050, Sacramento, California
  - Forest Investigative Site 034, Colorado Springs, Colorado
  - Forest Investigative Site 047, Cromwell, Connecticut
  - Forest Investigative Site 061, Gainesville, Florida
  - Forest Investigative Site 041, Orange City, Florida
  - Forest Investigative Site 059, Orlando, Florida
  - Forest Investigative Site 014, Spring Hill, Florida
  - Forest Investigative Site 055, West Palm Beach, Florida
  - Forest Investigative Site 058, Blue Ridge, Georgia
  - Forest Investigative Site 031, Savannah, Georgia
  - Forest Investigative Site 022, Chicago, Illinois
  - Forest Investigative Site 010, Peoria, Illinois
  - Forest Investigative Site 005, Indianapolis, Indiana
  - Forest Investigative Site 017, Louisville, Kentucky
  - Forest Investigative Site 009, Ann Arbor, Michigan
  - Forest Investigative Site 024, Rochester Hills, Michigan
  - Forest Investigative Site 036, Stevensville, Michigan
  - Forest Investigative Site 049, Whitehouse Station, New Jersey
  - Forest Investigative Site 018, Albuquerque, New Mexico
  - Forest Investigative Site 062, Raleigh, North Carolina
  - Forest Investigative Site 052, Winston-Salem, North Carolina
  - Forest Investigative Site 038, Akron, Ohio
  - Forest Investigative Site 016, Cincinnati, Ohio
  - Forest Investigative Site 015, Dayton, Ohio
  - Forest Investigative Site 019, Middleburg Heights, Ohio
  - Forest Investigative Site 001, Oklahoma City, Oklahoma
  - Forest Investigative Site 027, Oklahoma City, Oklahoma
  - Forest Investigative Site 066, Mechanicsburg, Pennsylvania
  - Forest Investigative Site 054, Philadelphia, Pennsylvania
  - Forest Investigative Site 046, Greer, South Carolina
  - Forest Investigative Site 023, Austin, Texas
  - Forest Investigative Site 003, San Antonio, Texas
  - Forest Investigative Site 042, San Antonio, Texas
  - Forest Investigative Site 025, Clinton, Utah
  - Forest Investigative Site 013, Salt Lake City, Utah
  - Forest Investigative Site 021, Lynchburg, Virginia
  - Forest Investigative Site 006, Bellevue, Washington
  - Forest Investigative Site 063, Seattle, Washington
  - Forest Investigative Site 004, Racine, Wisconsin

REFERENCES:
- [Derived] Arnold LM, Bateman L, Palmer RH, Lin Y. Preliminary experience using milnacipran in patients with juvenile fibromyalgia: lessons from a clinical trial program. Pediatr Rheumatol Online J. 2015 Jun 26;13:27. doi: 10.1186/s12969-015-0025-9. PMID 26112278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited over a 12 month period from April of 2011 to April of 2012 at 47 study sites in the United States.
Pre-assignment Details: 116 patients took at least 1 dose of open-label investigational product; 20 patients were randomized to receive double-blind treatment.
Groups:
- Milnacipran: Maximum tolerated dose (50, 75, or 100 mg/day tablets) was determined during the open-label phase of the study. Oral administration, twice daily dosing
Period: Open-Label Period
Arm/Group | Milnacipran | Placebo
Started | 116 | 0
Completed | 20 | 0
Not Completed | 96 | 0
Not completed — Inclusion/exclusion criteria not met | 66 | 0
Not completed — Adverse Event | 8 | 0
Not completed — Lack of Efficacy | 3 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 9 | 0
Not completed — Lost to Follow-up | 6 | 0
Not completed — Other Reason | 2 | 0
Period: Double-Blind Period
Arm/Group | Milnacipran | Placebo
Started | 14 | 6
Completed | 12 | 6
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: All demographic data was based on the Open-Label Safety Population, which consists of 116 patients who took at least 1 dose of open-label milnacipran.
Groups:
- Open-Label Milnacipran: Maximum tolerated dose (50, 75, or 100 mg/day tablets) determined during the open label treatment phase. Oral administration, twice daily dosing
Arm/Group | Open-Label Milnacipran
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (1.4)
Age, Customized [Number; unit: Participants]
  13 years old | 10
  14 years old | 21
  15 years old | 21
  16 years old | 23
  17 years old | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 18
Region of Enrollment [Number; unit: Participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: Time to First Loss of Therapeutic Response (LTR) Following Randomization to Milnacipran or Placebo.
Description: During the open-label period, 20 patients out of 116 enrolled had a reduction from baseline (Visit 2) of at least 50% in their pain, were classified as responders and were randomized (Visit 7). A Loss of Therapeutic Response was said to occur if, during the double-blind treatment period, any of the following occurred: • A worsening of fibromyalgia requiring an alternate treatment OR • An increase in 1-week mean of daily pain ratings (11-point numeric rating scale) to greater than 70% of Baseline (Visit 2) OR • Withdrawal from the study for any reason except withdrawals due to extenuating circumstances
Time Frame: Change from Visit 7 (Week 8) to Visit 10 (Week 16)
Population: The Open-Label Safety Population consists of 116 patients who took at least 1 dose of open-label milnacipran. 20 patients who were randomized to a treatment group (Randomized Population) took at least 1 dose of double-blind treatment (Double-blind Safety Population) and were analyzed as randomized (Double-blind Intent-to-Treat [ITT] Population).
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Placebo: Dose matched placebo, oral administration, twice daily dosing
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 6 | 14
Days | NA (NA) — No patients in the placebo arm experienced a loss of therapeutic effect during the double-blind study period. | 7.0 (1.4)

2. Secondary Outcome: Patient Global Impression of Severity (PGIS)
Description: The wording of the PGIS assessment was as follows: "Considering all aspects of your illness, how do you evaluate the severity of your fibromyalgia?" The possible responses to this question were 1. Normal, not at all ill 2. Borderline ill 3. Mildly ill 4. Moderately ill 5. Severely ill 6. Extremely ill
Time Frame: Change from Visit 7 (Week 8) to Visit 10 (Week 16)
Population: The Open-Label Safety Population consists of 116 patients who took at least 1 dose of open-label milnacipran. 20 patients were randomized to a treatment group (Randomized Population) took at least 1 dose of double-blind treatment (Double-blind Safety Population) and were analyzed as randomized (Double-blind Intent-to-Treat [ITT] Population).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 6 | 14
units on a scale | 0.5 (0.8) | 0.4 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected over a 17-month period from April, 2011 to September, 2012
Groups:
- Milnacipran - Open-Label Treatment Period: Maximum tolerated dose (50, 75, or 100 mg/day tablets) was determined during a four-week dose escalation period, and then continued at the maximum tolerated dose for an additional four weeks. Oral administration, twice daily dosing
- Placebo - Double Blind-Treatment: Dose matched placebo, oral administration, twice daily dosing
- Milnacipran - Double-Blind Treatment Period: Maximum tolerated dose (50, 75, or 100 mg/day tablets) was determined during the open-label phase of the study. Oral administration, twice daily dosing
Arm/Group | Milnacipran - Open-Label Treatment Period | Placebo - Double Blind-Treatment | Milnacipran - Double-Blind Treatment Period
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/6 | 1/14
Other Adverse Events (participants affected / at risk) | 62/116 | 4/6 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran - Open-Label Treatment Period (N=116) | Placebo - Double Blind-Treatment (N=6) | Milnacipran - Double-Blind Treatment Period (N=14)
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran - Open-Label Treatment Period (N=116) | Placebo - Double Blind-Treatment (N=6) | Milnacipran - Double-Blind Treatment Period (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 7 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Noncardiac chest pain (General disorders) | 1 | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0 | 2
Headache (Nervous system disorders) | 12 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 38 | 0 | 0
Vomiting (Gastrointestinal disorders) | 16 | 0 | 0
Dizziness (Nervous system disorders) | 10 | 0 | 0
Fatigue (General disorders) | 7 | 0 | 0
Hot flush (Vascular disorders) | 7 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, no firm conclusions about the use of milnacipran in pediatric patients for the treatment of primary fibromyalgia can be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.